CLINICAL TRIAL: NCT05028062
Title: Testing the Reward-Drinker Hypothesis of Naltrexone Using an Extended-Release Formulation
Brief Title: Naltrexone in AUD Reward Drinkers
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 849558
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder; Alcoholism
Keywords: XR-NTX; Naltrexone; Alcohol
MeSH Terms: conditions — Alcoholism | interventions — Injections, Intramuscular; Practice Management, Medical

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, parallel-group clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- XR-NTX 380 mg, intramuscular injection (Active Comparator): Subjects will receive an injection of XR-NTX 380 mg (4 mL) repeated once after 4 weeks.
  Interventions: Drug: XR-NTX 380 mg, intramuscular injection; Behavioral: Medical Management
- Inactive placebo intramuscular injection (Placebo Comparator): Subjects will receive a placebo injection repeated once after 4 weeks.
  Interventions: Behavioral: Medical Management; Drug: Placebo intramuscular injection

INTERVENTIONS:
Drug: XR-NTX 380 mg, intramuscular injection — Two doses of XR-NTX 380 mg, intramuscular injection.
  Other Names: Vivitrol naltrexone for extended-release injectable suspension
  Arms: XR-NTX 380 mg, intramuscular injection
Behavioral: Medical Management — All subjects will receive 8 weeks of medical management (Pettinati et al. 2004) will support subjects' efforts to reduce or stop their drinking. The study nurse makes direct recommendations for reducing drinking to sensible levels. The first session will use the brochure A Guide to Sensible Drinking (WHO 1996). Subsequent treatment sessions (15-25 minutes) will be conducted at each study visit, during which the nurse will perform an assessment of the subject's drinking, and make recommendations to follow until the next visit. Men will be advised to consume no more than 3 drinks 4 times per week; women will be advised to consume no more than 2 drinks 4 times per week.
Drug: Placebo intramuscular injection — Two doses of XR-NTX 380 mg, intramuscular injection.
  Other Names: Inactive placebo
  Arms: Inactive placebo intramuscular injection

SUMMARY:
This study is a phase IV, two-arm, randomized, double-blind, placebo-controlled study to assess whether individuals identified as primarily reward drinkers are significantly more likely to reduce heavy drinking if they receive XR-NTX than a matching placebo injection.

Study subjects will receive monthly injections of long-acting injectable naltrexone 380 mg (4 mL) or matching placebo. All subjects will also receive 4 sessions of Medical Management (MM). Post-treatment follow-up visits will be conducted at 4 weeks after the scheduled completion of treatment.

DETAILED DESCRIPTION:
Study eligibility is determined at an initial screening visit, which can be completed in a single day or divided over multiple days. Portions of the screening may occur by telephone or video conference. Participants are asked not to drink before this and at all study visits. At all study visits, study staff will check breath alcohol level using a breathalyzer. If the breath alcohol level is greater than 0.02% (which can result from a single standard drink), participants may not be able to complete the visit.

Screening Visit: The screening visit will determine whether the study is a good fit for participants. It take about three hours to complete.

* Participants will be asked to show legal photo ID and undergo a breathalyzer test to ensure that the breath alcohol level is below 0.02% to complete this visit. A reading test wil be given to evaluate participant's ability to understand the consent form and study assessment questionnaires.
* Once the informed consent is complete a study clinician will complete a medical history and perform a physical examination. Study staff will draw approximately 3 tablespoons of blood for standard laboratory tests. Participants will also be asked to provide a urine sample to conduct a urinalysis, drug screen, and a urine pregnancy test (only for for women of childbearing potential--i.e., who have not had a hysterectomy, bilateral removal of the ovaries, or a tubal ligation or is less than two years postmenopausal). We will not include women who are pregnant, breast-feeding.
* Eligible participants will be required to provide the names and contact information of one or two people (trusted friends or family members) who may serve as additional contacts to assist staff with locating participants for safety or other study-related reasons.
* Participants will be asked to complete 4 assessments of about psychological health and alcohol and drug use history.

First Study Drug Visit (Week 1): Staff will contact participants within 1 week after completing the screening visit to inform eligibility status and schedule the next study visit.

* This visit will take approximately one and one-half hours to complete.
* Participants will be asked to complete a breathalyzer test and study staff will measure weight and vital signs (blood pressure and heart rate).
* Woman of childbearing potential, will be asked to provide a urine sample for a pregnancy test.
* Participants will be asked to complete 11 assessments about psychological health and alcohol and drug use history.
* Staff will instruct participants how to use the interactive voice response (IVR) system via telephone. During the 8 weeks of the study, participants will be asked to call a toll-free phone number each day, between 5:00 and 8:00 p.m. to connect to the system. Access to the system via a touch-tone phone requires a study ID and a password. The system has prompts to answer questions about feelings and use of alcohol on the day of the call and the preceding day. It takes about 5 to 8 minutes to complete the daily interview. The IVR system will provide a reminder if a call has not been completed by 8:15 p.m.
* The first brief counseling session will last about 45 minutes. The study nurse will discuss a treatment goal either to drink less or become completely abstinent. The nurse will also encourage participants to consider ways to reduce or stop drinking, based upon the treatment goal.
* Participants will be assigned to receive an injection of study medication administered by the nurse, which will be either XR-NTX or placebo (an inactive substance). The decision as to which medication received will be random, like a flip of a coin. The XR-NTX or placebo will look the same. Neither participants nor any of the study personnel will know which medication is received. In an emergency, though, the study staff in charge of the study medication can be contacted for that information.
* At each visit, study staff will ask about any side effects or other adverse events.

Biweekly Visits (Weeks 2, 4, and 6): At each biweekly visit:

* The staff will check breath alcohol concentration (Breathalyzer), weight, and vital signs and ask about any side effects or other adverse events that were experienced.
* Participants will asked to complete 6 assessments about psychological health and alcohol and drug use history. These should take about 20 minutes to answer.
* Participants will receive brief counseling from the study clinician, which will last about 20 minutes.
* At week 4, woman of childbearing potential, will have another urine pregnancy test. If the urine permanency test is positive, staff will discontinue the medication and the participant will be referred to an obstetrician for care.
* At week 4 the study nurse will give the second injection of XR-NTX or a placebo (an inactive substance)
* Participants will continue to call and complete the toll-free IVR number nightly.

  4. Endpoint Visit (Week 8): At this visit:
* The staff will measure breath alcohol concentration (Breathalyzer), weight, and vital signs and asked about any side effects or other adverse events that may have experienced.
* The study staff will ask you to complete 11 assessments about your psychological health and your alcohol and drug use history. These should take about 45 minutes to complete.
* Study staff will draw 1 tablespoonful of blood for lab tests.
* Participants will receive brief counseling from the study clinician, which will last about 20 minutes.

Follow-up Visits (4 weeks after endpoint visit): At the follow-up visit (which will take about one hour), the study staff will:

* Check breath alcohol concentration (Breathalyzer), weight and vital signs.
* Draw 1 tablespoonful of blood for lab tests.
* Participants will be asked to complete 9 assessments about psychological health and alcohol and drug use history.
* Once participants have completed the study, they will have an option to receive a letter to inform them whether they received XR-NTX or placebo medication.

Early Termination Visit

• Participants who choose to withdraw from the study before participation is complete will be asked to return to the research center for a visit to allow staff to administer the end-of-study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Willing to provide signed, informed consent and commit to completing the study procedures
* Able to read at an 8th grade or higher level
* Current DSM-5 diagnosis of AUD
* Reports consuming 24+ standard drinks (men) or 18+ standard drinks (women) weekly on average over the month prior to consent
* Expresses a desire to reduce or stop drinking and a willingness to receive two injections of study medication over 8 weeks of treatment.
* Either a reward drinker [i.e., an individual with a score of 19 or greater on the reward subscale and less than or equal to 18 on the relief subscale of the Inventory of Drinking Situations (IDS)] or a relief drinker (i.e., an individual with a score of 21 or greater on the relief subscale and less than or equal to 18 on the reward subscale of the IDS).
* Has a stable address in the local area; not planning to move; has documents for an ID check
* Women of child-bearing potential (i.e., who have not had a hysterectomy, bilateral oophorectomy, tubal ligation or are less than two years postmenopausal): must be non-lactating and practicing a reliable method of birth control and have a negative urine pregnancy test prior to the initiation of the study procedures. Examples of medically acceptable methods for this protocol include oral contraceptive pills, intrauterine device, injection of Depo-Provera, Norplant, contraceptive patch, contraceptive ring, double-barrier methods (such as condoms and diaphragm/spermicide), male partner sterilization, abstinence (and agreement to continue abstinence or to use an acceptable method of contraception, as listed above, should sexual activity commence).

Exclusion Criteria:

* Planned surgery within the timeframe of the study
* A current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation that could interfere with study participation or make it hazardous for the subject to do so (e.g., bleeding disorder, pancreatitis, epilepsy, diabetes, liver disease, kidney disease, or cardiomyopathy as determined by history and clinical exam); ALAT or ASAT concentration greater than 3 times the upper limit of normal (ULN), or direct bilirubin above the ULN. (Note-abnormal laboratory tests during screening may be repeated once).
* Chronic or episodic painful conditions that could require opioid medications for pain control
* History of seizure disorder (excluding childhood febrile seizures)
* History of allergy or other serious adverse event due to treatment with XR-NTX
* Current psychotic disorder (bipolar, schizophrenia, major depression with suicidal ideation, or psychotic features) identified by clinical examination or the structured interview that could interfere with study participation or make it hazardous for the subject.
* Current DSM-5 diagnosis of any drug use disorder other than alcohol, nicotine, or cannabis or a urine drug screen that is positive for benzodiazepines, opioids, amphetamines, cocaine or barbiturates.
* Current treatment with a psychotropic, anticonvulsant, opioid, anticoagulant or AUD treatment medication (i.e., naltrexone, acamprosate, disulfiram, topiramate, gabapentin, varenicline, or baclofen)
* Receipt of any experimental medication within the past 30 days
* In need of medical detoxification from alcohol
* Subjects cannot have been mandated by court for alcohol or drug abuse treatment or have pending legal proceedings that could result in incarceration within 6 months of enrollment.
* Homicidal or other behavioral disturbance that requires immediate clinical attention
* Judged by the principal investigator or his designee to be an unsuitable candidate for study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Frequency of heavy drinking days by medication group (timeline follow back calendar). | 8 weeks
  The number of Heavy Drinking Days during 8 weeks of treatment in the Naltrexone and placebo groups.

SECONDARY OUTCOMES:
Frequency of drinking days, and drinks/drinking day by medication group (timeline follow back calendar). | 8 weeks
  The number of Drinking Days, drinks/drinking day by medication group during 8 weeks of treatment in the Naltrexone and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Henry R Kranzler, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Studies of Addiction, Philadelphia, Pennsylvania, United States